CLINICAL TRIAL: NCT03984890
Title: Effect of Vitamin D3 Supplementation on Chronic Granulomatous Disease Patients With BCGosis/Itis
Brief Title: Vitamin D3 For CGD Patients With BCGosis/Itis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Jinqiao Sun, Professor, Children's Hospital of Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VDBCG
Record Dates: First submitted 2018-12-05; First posted 2019-06-13 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Vitamin D3; Chronic-granulomatous Disease; BCG
MeSH Terms: conditions — Granulomatous Disease, Chronic | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D Group (Experimental): Vitamin D3 Supplementation plus traditional treatment of CGD and TB
  Interventions: Drug: Vitamin D3; Drug: Traditional treatment of CGD and TB
- Control Group (Other): Traditional treatment of CGD and TB without Vitamin D Supplementation
  Interventions: Drug: Traditional treatment of CGD and TB

INTERVENTIONS:
Drug: Vitamin D3 — Vitamin D3 drops 800IU/d for 3 months
  Arms: Vitamin D Group
Drug: Traditional treatment of CGD and TB — Anti-tuberculosis drugs, interferon-gamma

SUMMARY:
When children with chronic granulomatous disease (CGD) got BCG infection the treatment would be a tough task. The goal of the proposed research is to observe weather vitamin D supplementation can help the CGD children get through this challenge.

DETAILED DESCRIPTION:
Chronic granulomatous disease (CGD) is one of primary immunodeficiency diseases. Due to the deficiency of the phagocyte nicotinamide adenine dinucleotide phosphate (NADPH) oxidase the respiratory burst of all types of phagocytic cells is badly impaired which lead to a susceptibility to infection among CGD patients.

BCG vaccine is wildly used in China to avoid severe tuberculosis infection. Children are supposed to get BCG vaccine injected within 24 hours after birth. When patients with CGD got the vaccination of BCG they will easily got infected. And due to the immunodeficiency of these children, the infection cannot be cure by normal treatment.

Vitamin D supplementation was used to treat tuberculosis in the pre-antibiotic era and is reported to have influence on immune system especially on monocytes and macrophages thus may help CGD children defend the BCG infection. In addition, studies show that 1,25-Dihydroxyvitamin D3 can induce nitric oxide synthase thus may up regulate NO production and help host defense against human tuberculosis without the help of NADPH oxidase. Other researches indicate that Vitamin D and the expression of vitamin D receptor may lead to induction of antimicrobial peptide such as LL-37 which help macrophages kill the intracellular Mycobacterium tuberculosis. These discoveries indicated that vitamin D may induce immune response against BCG in a nontraditional way. Therefore, when CGD patients face BCG infection, add vitamin D supplementation to the treatment may help them survive this challenge.

Since there have had clinical trials revealing that intermittent high dose vitamin D3 supplementation as 2.5mg per 14 days only receive positive effect on partial patients the investigators decide to choose a mild dose treatment as 800IU/d for 3 month to see if things get different in this way.

ELIGIBILITY:
Inclusion Criteria:

1. less than 18 years' old
2. Diagnosed with CGD
3. Got BCG infection after vaccination

Exclusion Criteria:

1. Serum 25-(OH)-vit D >75 nmol/L (30 ng/mL)
2. Hyperphosphatemia
3. Hypercalcemia
4. Acute or chronic renal failure
5. Acute or chronic cardiac failure
6. Kidney stone

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Mortality | 8 weeks
  Death rate among patients
Rate of Sputum Culture acid-fast bacilli microscopy Conversion | 8 weeks
  If sputum culture and acid-fast bacilli microscopy show positive results before treatments, compare the results before and after treatments to see if the rate that results changed from positive to negative differ between control group and vitamin D group
Duration of Fever | 8 weeks
  Calculate the days suffer from fevers to show the severity of the infection and the efficacy of the treatment
Number of Anti-tuberculosis Drugs Used in the Treatment | 8 weeks
  Calculate the number of anti-tuberculosis drugs used in the treatment to show the severity of the infection and the efficacy of the treatment
Urine Protein | 8 weeks
  Urine protein quantitation
Urine Calcium | 8 weeks
  Concentration of calcium in urine
Serum Levels of 25-OH Vitamin D3 | 8 weeks
  Concentration of 25-OH Vitamin D3 in serum
Serum Levels of Calcium | 8 weeks
  Concentration of calcium in serum

SECONDARY OUTCOMES:
Change in BMI | 1 year
  Evaluate the change in BMI by calculating weight(kg)/height(m)^2 before treatment and 1year after the treatment
Frequency of Recurrent Infections | 1 year
  Use frequency of recurrent infections to evaluate long-term benefits

CONTACTS AND LOCATIONS:
Overall Officials: Weili Yan, Ph.D, Study Director — Children's Hospital of Fudan University
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martineau AR, Wilkinson KA, Newton SM, Floto RA, Norman AW, Skolimowska K, Davidson RN, Sorensen OE, Kampmann B, Griffiths CJ, Wilkinson RJ. IFN-gamma- and TNF-independent vitamin D-inducible human suppression of mycobacteria: the role of cathelicidin LL-37. J Immunol. 2007 Jun 1;178(11):7190-8. doi: 10.4049/jimmunol.178.11.7190. PMID 17513768
- [Background] Rockett KA, Brookes R, Udalova I, Vidal V, Hill AV, Kwiatkowski D. 1,25-Dihydroxyvitamin D3 induces nitric oxide synthase and suppresses growth of Mycobacterium tuberculosis in a human macrophage-like cell line. Infect Immun. 1998 Nov;66(11):5314-21. doi: 10.1128/IAI.66.11.5314-5321.1998. PMID 9784538
- [Background] Martineau AR, Timms PM, Bothamley GH, Hanifa Y, Islam K, Claxton AP, Packe GE, Moore-Gillon JC, Darmalingam M, Davidson RN, Milburn HJ, Baker LV, Barker RD, Woodward NJ, Venton TR, Barnes KE, Mullett CJ, Coussens AK, Rutterford CM, Mein CA, Davies GR, Wilkinson RJ, Nikolayevskyy V, Drobniewski FA, Eldridge SM, Griffiths CJ. High-dose vitamin D(3) during intensive-phase antimicrobial treatment of pulmonary tuberculosis: a double-blind randomised controlled trial. Lancet. 2011 Jan 15;377(9761):242-50. doi: 10.1016/S0140-6736(10)61889-2. Epub 2011 Jan 5. PMID 21215445
- [Background] Liu PT, Stenger S, Li H, Wenzel L, Tan BH, Krutzik SR, Ochoa MT, Schauber J, Wu K, Meinken C, Kamen DL, Wagner M, Bals R, Steinmeyer A, Zugel U, Gallo RL, Eisenberg D, Hewison M, Hollis BW, Adams JS, Bloom BR, Modlin RL. Toll-like receptor triggering of a vitamin D-mediated human antimicrobial response. Science. 2006 Mar 24;311(5768):1770-3. doi: 10.1126/science.1123933. Epub 2006 Feb 23. PMID 16497887
- [Background] Collaborative Group for the Meta-Analysis of Individual Patient Data in MDR-TB treatment-2017; Ahmad N, Ahuja SD, Akkerman OW, Alffenaar JC, Anderson LF, Baghaei P, Bang D, Barry PM, Bastos ML, Behera D, Benedetti A, Bisson GP, Boeree MJ, Bonnet M, Brode SK, Brust JCM, Cai Y, Caumes E, Cegielski JP, Centis R, Chan PC, Chan ED, Chang KC, Charles M, Cirule A, Dalcolmo MP, D'Ambrosio L, de Vries G, Dheda K, Esmail A, Flood J, Fox GJ, Frechet-Jachym M, Fregona G, Gayoso R, Gegia M, Gler MT, Gu S, Guglielmetti L, Holtz TH, Hughes J, Isaakidis P, Jarlsberg L, Kempker RR, Keshavjee S, Khan FA, Kipiani M, Koenig SP, Koh WJ, Kritski A, Kuksa L, Kvasnovsky CL, Kwak N, Lan Z, Lange C, Laniado-Laborin R, Lee M, Leimane V, Leung CC, Leung EC, Li PZ, Lowenthal P, Maciel EL, Marks SM, Mase S, Mbuagbaw L, Migliori GB, Milanov V, Miller AC, Mitnick CD, Modongo C, Mohr E, Monedero I, Nahid P, Ndjeka N, O'Donnell MR, Padayatchi N, Palmero D, Pape JW, Podewils LJ, Reynolds I, Riekstina V, Robert J, Rodriguez M, Seaworth B, Seung KJ, Schnippel K, Shim TS, Singla R, Smith SE, Sotgiu G, Sukhbaatar G, Tabarsi P, Tiberi S, Trajman A, Trieu L, Udwadia ZF, van der Werf TS, Veziris N, Viiklepp P, Vilbrun SC, Walsh K, Westenhouse J, Yew WW, Yim JJ, Zetola NM, Zignol M, Menzies D. Treatment correlates of successful outcomes in pulmonary multidrug-resistant tuberculosis: an individual patient data meta-analysis. Lancet. 2018 Sep 8;392(10150):821-834. doi: 10.1016/S0140-6736(18)31644-1. PMID 30215381